CLINICAL TRIAL: NCT01150994
Title: Emergency Department Safety Assessment and Follow-up Evaluation (ED-SAFE)
Acronym: ED-SAFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Edwin Boudreaux, Study Principal Investigator, University of Massachusetts, Worcester
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Screening
Other Study IDs: 13420; 1U01MH088278-01 (NIH)
Record Dates: First submitted 2010-06-24; First posted 2010-06-25 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Suicide
Keywords: Suicide screening among ED patients
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Treatment as Usual (No Intervention)
- Screening Alone (No Intervention): Enhanced screening among ED patients
- Safety Assessment and Follow-up Telephone Intervention (Experimental): SAFTI: Safety Assessment in the ED combine with a Follow-up Telephone Intervention.
  Interventions: Behavioral: Safety Assessment and Follow-up Telephone Intervention (SAFTI).

INTERVENTIONS:
Behavioral: Safety Assessment and Follow-up Telephone Intervention (SAFTI). — Mental health evaluation in ED, followed by Post-ED counseling
  Arms: Safety Assessment and Follow-up Telephone Intervention

SUMMARY:
The NIMH s RFA-Suicide Prevention in Emergency Medicine Departments recognizes the emergency department (ED) as an important setting to increase suicide detection and prevention efforts but observes that evidence-based practice guidelines do not exist. In response, we have designed the Emergency Department Safety Assessment and Follow-up Evaluation (ED-SAFE) trial. The ED-SAFE study will be conducted using a quasi-experimental design appropriate for studying systems-based change. The study consists of two components (Screening Outcome & Intervention Evaluation) and three phases of data collection: Treatment as Usual, Screening Alone, and Intervention. During each phase, 480 suicidal patients (1,440 total) will be enrolled and followed using multiple methods for 12 months.

The Screening Outcome Component

The Screening Outcome component will use data collected during the Treatment as Usual and Screening Alone phases. Consistent with systems-change principles, when universal screening is incorporated during the Screening Alone phase, it will be completed by the primary nurse as part of routine care. Primarily, it will focus on testing a practical approach to screen ED patients for suicidal ideation and behavior and will assess its impact on suicide detection, process outcomes, and suicide behaviors.

Intervention Evaluation Component

The Intervention Evaluation component will use data from the Treatment as Usual, Screening Alone, and Intervention Phases. During the Intervention phase, each ED will implement a multi-component, systems-based Intervention called the Safety Assessment and Follow-up Telephone Intervention (SAFTI). The SAFTI will combine elements of: (a) safety planning administered by nursing staff in the ED, and (b) Coping Long Term with Active Suicide Program (CLASP)-ED, a series of up to 7 semi-structured telephone advising calls to the patient and 4 to the significant other over the 12 months after the ED visit. Safety planning will be implemented universally to all suicidal patients, regardless of whether they are ultimately enrolled into the trial, as part of a comprehensive suicide management protocol (e.g., it is a systems-based change). However, for practical and budgetary considerations, the CLASP-ED telephone advising calls will be administered only to participants enrolled into the study.

Our overarching hypotheses will be tested using a combination of the Screening Outcome component and the Intervention Evaluation Component. We predict that screening will improve detection of suicidal ideation, and the intervention will enhance the quality of care and reduce suicide outcomes.

DETAILED DESCRIPTION:
see summary above

ELIGIBILITY:
Inclusion Criteria:

* Over 18,
* Entering care at a hospital ED,
* Documented thoughts or behaviors related to self-harm.

Exclusion Criteria:

* No phone or permanent address,
* Does not speak English or Spanish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1440 (Actual)
Dates: Start 2010-07; Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Percentage of ER patients screened for self harm | July 2010 - November 2013
Quality of care | July 2010 - November 2014
  * Process outcomes (e.g. receipt of safety plan)
  * Involvement in behavioral health treatment
Suicide-related outcomes | July 2010 - November 2014
  * Preparatory acts
  * Suicide attempts
  * Completed suicides

CONTACTS AND LOCATIONS:
Overall Officials: Edwin Boudreaux, PhD, Principal Investigator — UMass Medical School; Carlos Camargo, MD, DrPH, Principal Investigator — Massachusetts General Hospital; Ivan Miller III, PhD, Principal Investigator — Butler Hospital
Locations (8):
- United States (8):
  - Maricopa Medical Center, Phoenix, Arizona
  - University of Arkansas Medical Center, Little Rock, Arkansas
  - University of Colorado Hospital, Aurora, Colorado
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - UMass Medical School, Marlborough Hospital, Worcester, Massachusetts
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Ohio State University Medical Center, Columbus, Ohio
  - Memorial Hospital of Rhode Island, Pawtucket, Rhode Island

REFERENCES:
- [Result] Arias SA, Zhang Z, Hillerns C, Sullivan AF, Boudreaux ED, Miller I, Camargo CA. Using structured telephone follow-up assessments to improve suicide-related adverse event detection. Suicide Life Threat Behav. 2014 Oct;44(5):537-47. doi: 10.1111/sltb.12088. Epub 2014 Mar 3. PMID 24588679
- [Result] Betz ME, Sullivan AF, Manton AP, Espinola JA, Miller I, Camargo CA Jr, Boudreaux ED; ED-SAFE Investigators. Knowledge, attitudes, and practices of emergency department providers in the care of suicidal patients. Depress Anxiety. 2013 Oct;30(10):1005-12. doi: 10.1002/da.22071. Epub 2013 Feb 20. PMID 23426881
- [Result] Betz ME, Miller M, Barber C, Miller I, Sullivan AF, Camargo CA Jr, Boudreaux ED; ED-SAFE Investigators. Lethal means restriction for suicide prevention: beliefs and behaviors of emergency department providers. Depress Anxiety. 2013 Oct;30(10):1013-20. doi: 10.1002/da.22075. Epub 2013 Mar 14. PMID 23495002
- [Result] Betz ME, Arias SA, Miller M, Barber C, Espinola JA, Sullivan AF, Manton AP, Miller I, Camargo CA Jr, Boudreaux ED. Change in emergency department providers' beliefs and practices after use of new protocols for suicidal patients. Psychiatr Serv. 2015 Jun;66(6):625-31. doi: 10.1176/appi.ps.201400244. Epub 2015 Mar 1. PMID 25726978
- [Result] Boudreaux ED, Miller I, Goldstein AB, Sullivan AF, Allen MH, Manton AP, Arias SA, Camargo CA Jr. The Emergency Department Safety Assessment and Follow-up Evaluation (ED-SAFE): method and design considerations. Contemp Clin Trials. 2013 Sep;36(1):14-24. doi: 10.1016/j.cct.2013.05.008. Epub 2013 May 22. PMID 23707435
- [Result] Caterino JM, Sullivan AF, Betz ME, Espinola JA, Miller I, Camargo CA Jr, Boudreaux ED; Emergency Department Safety Assessment and Follow-up Evaluation (ED-SAFE) Investigators. Evaluating current patterns of assessment for self-harm in emergency departments: a multicenter study. Acad Emerg Med. 2013 Aug;20(8):807-15. doi: 10.1111/acem.12188. PMID 24033624
- [Result] Ting SA, Sullivan AF, Boudreaux ED, Miller I, Camargo CA Jr. Trends in US emergency department visits for attempted suicide and self-inflicted injury, 1993-2008. Gen Hosp Psychiatry. 2012 Sep-Oct;34(5):557-65. doi: 10.1016/j.genhosppsych.2012.03.020. Epub 2012 May 2. PMID 22554432
- [Result] Ting SA, Sullivan AF, Miller I, Espinola JA, Allen MH, Camargo CA Jr, Boudreaux ED; Emergency Department Safety and Follow-up Evaluation (ED-SAFE) Investigators. Multicenter study of predictors of suicide screening in emergency departments. Acad Emerg Med. 2012 Feb;19(2):239-43. doi: 10.1111/j.1553-2712.2011.01272.x. Epub 2012 Jan 30. PMID 22288721
- [Derived] Brown LA, Boudreaux ED, Arias SA, Miller IW, May AM, Camargo CA Jr, Bryan CJ, Armey MF. C-SSRS performance in emergency department patients at high risk for suicide. Suicide Life Threat Behav. 2020 Dec;50(6):1097-1104. doi: 10.1111/sltb.12657. Epub 2020 Jul 24. PMID 32706437
- [Derived] Boudreaux ED, Camargo CA Jr, Arias SA, Sullivan AF, Allen MH, Goldstein AB, Manton AP, Espinola JA, Miller IW. Improving Suicide Risk Screening and Detection in the Emergency Department. Am J Prev Med. 2016 Apr;50(4):445-453. doi: 10.1016/j.amepre.2015.09.029. Epub 2015 Dec 4. PMID 26654691